CLINICAL TRIAL: NCT00696852
Title: Effects of Mindfulness and Yoga on Heart Rate Variability and Immune Markers
Brief Title: Mindfulness, Yoga, and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joan Fox, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHBI-1201
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Cardiovascular Disease; Stress; Anxiety; Depression
Keywords: Mindfulness; Meditation; Yoga; Inflammatory Markers
MeSH Terms: conditions — Cardiovascular Diseases; Anxiety Disorders; Depression | interventions — Mindfulness; Yoga; Exercise; Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness Meditation (Active Comparator)
  Interventions: Behavioral: Mindfulness Meditation
- Yoga (Active Comparator)
  Interventions: Behavioral: Yoga
- Conventional Stress Reduction (Active Comparator)
  Interventions: Behavioral: Exercise, Relaxation, and Health Education

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The yoga and mindfulness classes will combine specific techniques of meditation, simple yoga postures, and breathing exercises.
  Other Names: MBSR
  Arms: Mindfulness Meditation
Behavioral: Yoga — The yoga and mindfulness classes will combine specific techniques of meditation, simple yoga postures, and breathing exercises.
  Arms: Yoga
Behavioral: Exercise, Relaxation, and Health Education — The Exercise, Relaxation and Health Education program will consist of a 90 min group session that will include simple relaxation (such as progressive muscle relaxation) and light stretching exercises, group support, and discussions of various health topics and on stress reduction.
  Other Names: Progressive muscle relaxation
  Arms: Conventional Stress Reduction

SUMMARY:
In this study, we will conduct a preliminary, yet comprehensive evaluation of Mindfulness and Yoga, as compared to an exercise and education-based stress-reduction program. and simultaneous evaluation of the effect of an 8 week program of Mindfulness, 12 weeks of Yoga practice, and 12 weeks of an exercise and education-based program.

105 otherwise healthy individuals, who have cardiovascular risk factors and mild to moderate stress or anxiety will be randomly assigned to one of the three intervention groups: an 8 week program of Mindfulness, 12 week program of Yoga practice, and 12 week exercise and education-based group program. All subjects will perform daily practice that will continue after the weekly sessions end, allowing a follow up assessment at 24 weeks. Self-reported mood and psychological distress and physiological indicators of function of the ANS and stress hormones will be assessed at baseline, 8 weeks, 12 weeks and 24 weeks. Blood and urine samples will be collected at baseline and 8 weeks to determine levels inflammatory and atherosclerosis markers.

We anticipate that the study will provide information on the efficacy of the Mindfulness and Yoga interventions as stress-reduction practices, variability in potential markers for activation of the brain/cardiovascular system connections, and preliminary estimates of effect size for each of these markers. Thus, the study will provide the data needed for designing a future study that will rigorously address these questions in a larger, randomized trial of Mindfulness and Yoga in patients with cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 40 and 75
* A Framingham score >10
* A DASS-21 anxiety score >5
* A DASS-21 stress score >10
* A DASS-21 depression score > than 6
* A systolic blood pressure > 140
* A diastolic blood pressure > 90
* Diagnosed with diabetes
* Willing to accept randomization into and participation in one of the three intervention programs: Mindfulness, Yoga, or Conventional Stress Reduction

Exclusion Criteria:

* Already practicing Mindfulness, Yoga, or similar meditative mind-body practices on a weekly basis
* Already enrolled in a lifestyle modification program including exercise or diet program
* Yoga or meditation be incompatible with religious or philosophical beliefs
* Experienced a major stressful life event in the last three months prior to the beginning of the intervention that is likely to affect the outcomes of the study
* Currently being treated or on medications for psychiatric conditions, including depression, anxiety, anger, or hostility
* A depression score >20 on the DASS-21 questionnaire
* A history of myocardial disease, peripheral vascular disease, cerebrovascular disease, atrial fibrillation, pacemaker placement, heart failure, valvular heart disease, congenital heart disease, Wolf-Parkinson White Syndrome, cardiomyopathy, or severe left ventricular systolic dysfunction
* Take melatonin supplements or any herbal supplement that contains melatonin or 5-LO inhibitors (turmeric, curcumin, ginger and frankincense herbal extracts)
* Currently using any drugs that contain beta-adrenergic blocking agents, beta-agonists, glucocorticoids, psychotropic medications, drugs that block 5-LO pathway (zileuton, monetlukast), TNF-a blocking agents (infliximab, etanercept, adalimumab)
* A planned change in blood pressure, anticoagulant medication and lipids lower agents (such as aspirin, statin and plavix) 1 month prior and during the intervention
* Asthma, obstructive pulmonary disease, or any other respiratory disease
* Pregnant or breastfeeding
* An active/chronic infection, cancer, connective tissue, or other inflammatory disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
change in inflammatory markers | within 26 weeks of enrollment

SECONDARY OUTCOMES:
change in psychological and physiological markers of anxiety, depression, and cardiovascular disease | within 26 weeks from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joan EB Fox, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States